CLINICAL TRIAL: NCT02442388
Title: Postoperative Pain of Root Canal Therapy With Three Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Shokraneh, DDS, MS, AssistantProfessor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9308
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Pain
Keywords: pain; root canal therapy; endodontics; file
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hand file (Experimental): Instrumentation technique
  Interventions: Procedure: Instrumentation technique with hand file
- ProTaper file (Experimental): Instrumentation technique
  Interventions: Procedure: Instrumentation technique with ProTaper
- Wave-One file (Experimental): Instrumentation technique
  Interventions: Procedure: Instrumentation technique with WaveOne

INTERVENTIONS:
Procedure: Instrumentation technique with hand file — type of instrumentation technique for root canal treatment
  Arms: Hand file
Procedure: Instrumentation technique with ProTaper — type of instrumentation technique for root canal treatment
  Arms: ProTaper file
Procedure: Instrumentation technique with WaveOne — type of instrumentation technique for root canal treatment
  Arms: Wave-One file

SUMMARY:
The purpose of this prospective, randomized, double-blind study was to compare the prospective pain in asymptomatic mandibular molar teeth with necrotic pulp and periapical lesion using three different instrumentation files: Hand, Protaper Universal, and Wave-One files.

DETAILED DESCRIPTION:
ProTaper Universal system is one of the conventional multi-file rotary systems that prepared root canals with six files: three shaping files and three finishing files. A unique design element is varying tapers along the instruments' long axes. The three shaping files have tapers that increase coronally, and the reverse pattern is seen in the five finishing files. Wave-One is reciprocation-based systems that instrumented root canals with only single file. Some studies demonstrated that it has outperformed conventional continuous rotary nickel-titanium (NiTi) preparation in some aspects. The reciprocating motion of Wave-One relieves the stress on the file by special counterclockwise (cutting action) and clockwise (release of the instrument) movements and, therefore, extends the durability of a NiTi instrument and increases its fatigue resistance in comparison with continuous rotation motion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient

Exclusion Criteria:

* Allergy to anesthetics, pregnancy, breastfeeding, vital teeth, unrestorable teeth, and teeth associated with pain or swelling

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain as assessed by Heft-Parker VAS | After each technique, up to 72 hours
  Pain as assessed by Heft-Parker VAS